CLINICAL TRIAL: NCT04578756
Title: A 52-Week, Multicenter, Open-Label, Flexible-dose Study to Evaluate the Long-term Safety and Tolerability of Cariprazine in the Treatment of Pediatric Subjects With Schizophrenia, Bipolar I Disorder, or Autism Spectrum Disorder
Brief Title: Open-Label, Flexible-dose Study to Evaluate the Long-Term Safety and Tolerability of Cariprazine in the Treatment of Pediatric Participants With Schizophrenia, Bipolar I Disorder, or Autism Spectrum Disorder
Acronym: 3070 Ped OLE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3070-301-001
Record Dates: First submitted 2020-10-01; First posted 2020-10-08 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Schizophrenia; Bipolar I Disorder; Autism Spectrum Disorder (ASD)
Keywords: Schizophrenia; Bipolar I Disorder; Cariprazine; Autism Spectrum Disorder (ASD)
MeSH Terms: conditions — Schizophrenia; Autism Spectrum Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (11):
- Cariprazine Dose 1 (Experimental): Participants with Schizophrenia (age 13 to 17 years and < 40 kg body weight) will receive cariprazine.
  Interventions: Drug: Cariprazine Flexible Dose
- Cariprazine Dose 2 (Experimental): Participants with Schizophrenia (age 13 to 17 years and >= 40 kg body weight) will receive cariprazine.
  Interventions: Drug: Cariprazine Flexible Dose
- Cariprazine Dose 3 (Experimental): Participants with Bipolar I Disorder (age 10 to 12 years and <40 kg body weight) will receive cariprazine.
  Interventions: Drug: Cariprazine Flexible Dose
- Cariprazine Dose 4 (Experimental): Participants with Bipolar I Disorder (age 10 to 12 years and >= 40 kg body weight) will receive cariprazine.
  Interventions: Drug: Cariprazine Flexible Dose
- Cariprazine Dose 5 (Experimental): Participants with Bipolar I Disorder (age 13 to 17 years and < 40 kg body weight) will receive cariprazine.
  Interventions: Drug: Cariprazine Flexible Dose
- Cariprazine Dose 6 (Experimental): Participants with Bipolar I Disorder (age 13 to 17 years and >= 40 kg body weight) will receive cariprazine.
  Interventions: Drug: Cariprazine Flexible Dose
- Cariprazine Dose 7 (Experimental): Participants with Autism Spectrum Disorder ( age 5 to 9 years) will receive cariprazine.
  Interventions: Drug: Cariprazine Flexible Dose
- Cariprazine Dose 8 (Experimental): Participants with Autism Spectrum Disorder (age 10 to 12 years and <40 kg weight) will receive cariprazine.
  Interventions: Drug: Cariprazine Flexible Dose
- Cariprazine Dose 9 (Experimental): Participants with Autism Spectrum Disorder (age 10 to 12 years and >=40 kg body weight) will receive cariprazine.
  Interventions: Drug: Cariprazine Flexible Dose
- Cariprazine Dose 10 (Experimental): Participants with Autism Spectrum Disorder (age 13 to 17 years and <40 kg weight) will receive cariprazine.
  Interventions: Drug: Cariprazine Flexible Dose
- Cariprazine Dose 11 (Experimental): Participants with Autism Spectrum Disorder (age 13 to 17 years and >= 40 kg body weight) will receive cariprazine.
  Interventions: Drug: Cariprazine Flexible Dose

INTERVENTIONS:
Drug: Cariprazine Flexible Dose — 1 capsule to be taken orally at approximately the same time of day (morning or evening)
  Arms: Cariprazine Dose 1; Cariprazine Dose 10; Cariprazine Dose 11; Cariprazine Dose 2; Cariprazine Dose 3; Cariprazine Dose 4; Cariprazine Dose 5; Cariprazine Dose 6; Cariprazine Dose 8; Cariprazine Dose 9
Drug: Cariprazine Flexible Dose — Dose solution (in milliliters) to be taken orally at approximately the same time of day (morning or evening)
  Arms: Cariprazine Dose 7

SUMMARY:
The purpose of this study is to evaluate the long-term safety and tolerability of cariprazine in the treatment of pediatric participants with schizophrenia, bipolar I disorder, or autism spectrum disorder (ASD) and to establish the benefit-risk profile of long-term treatment in this population.

ELIGIBILITY:
Inclusion Criteria:

* Participants with Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition Text Revision (DSM-5-TR) primary diagnosis of schizophrenia or bipolar I disorder, or autism spectrum disorder as confirmed by Kiddie Schedule for Affective Disorders and Schizophrenia for School-Age Children-Present and Lifetime Version (K-SADS-PL) at the Screening Visit 1 (for de novo subjects, or as previously confirmed in parent study for subjects who completed Study 3112-301-001 or M21-465).
* De novo participants must have normal physical examination findings, clinical laboratory test results, and electrocardiogram (ECG) results at Screening Visit 1. Abnormal results must not be clinically significant as determined by the investigator. Participants enrolling after completion of Study M21-465 or 3112-301-001 have had monitoring of laboratory tests, physical examinations, and ECGs at the completion visit of the parent studies.
* Participant must have a caregiver (parent or legally authorized representative) who is willing and able to be responsible for safety monitoring of the participant, provide information about the participant's condition, oversee administration of study intervention, and accompany the participant to all study visits.

Exclusion Criteria:

* Participants with DSM-5-TR diagnosis of major depressive disorder, schizoaffective disorder, schizophreniform disorder, brief psychotic disorder, or psychotic disorder due to another medical condition. Participants with ASD that is associated with Rett disorder, fragile-X syndrome, or childhood disintegrative disorder.
* Prior DSM-5-TR diagnosis of intellectual disability (IQ < 70) for schizophrenia and bipolar I disorder participants. Prior DSM-5-TR diagnosis of profound intellectual disability (IQ < 25) for ASD participants.
* Participant has a condition or is in a situation, which, in the investigator's opinion, may put the participant at significant risk, may confound the study results, or may interfere significantly with the participant's participation in the study.

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 310 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2025-10-06 (Actual); Study Completion 2025-10-06 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Treatment-emergent Adverse Events (TEAEs) in the Treatment Period | Baseline Day 1 to Week 59
  An adverse event (AE) is any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. An adverse event can therefore be any unfavorable and unintended sign (i.e. laboratory value), symptom, or disease temporally associated with the use of a medicinal product, whether or not related to the medicinal product. A TEAE is an AE that occurs or worsens after receiving study drug.
Number of Participants With Clinically Significant Changes From Baseline in Clinical Laboratory Parameters | Baseline Day 1 to Week 52
  Clinical laboratory parameters included tests of hematology, chemistry, urinalysis and prolactin. The investigator assessed the results for clinical significance.
Number of Participants With Clinically Significant Changes From Baseline in Vital Sign Parameters | Baseline Day 1 to Week 59
  Vital sign parameters included blood pressure, pulse rate, body mass index (BMI), weight, and waist circumference. The investigator assessed the results for clinical significance.
Number of Participants With Clinically Significant Changes From Baseline in Electrocardiograms (ECG) | Baseline Day 1 to Week 52
  A standard 12-lead ECG was performed. The investigator determined the clinical significance of the ECG findings using the central ECG interpretation laboratory report.
Number of Participants With Suicidal Ideation or Suicidal Behavior as Recorded on the Columbia-Suicide Severity Rating (C-SSRS) Scale | Baseline Day 1 to Week 52
  C-SSRS is a clinician-rated scale that reports the severity of both suicidal ideation and behavior. Suicidal ideation is classified on a 5-item scale: 1 "wish to be dead," and 5 "active suicidal ideation with specific plan and intent". Suicidal behavior is classified on a 5-item scale: 0 "no suicidal behavior, and 4 "actual attempt".
Change From Baseline in Abnormal Involuntary Movement Scale (AIMS) | Baseline Day 1 to Week 52
  AIMS assesses abnormal involuntary movements, such as tardive dyskinesia, associated with antipsychotic drugs; it measures facial, oral, extremities, and trunk movements, as well as the participant's awareness of abnormal movements. The first 10 items are rated on a none (0) to severe (4) scale. There are an additional 2 items on dental status that are answered yes or no.
Change From Baseline in Barnes Akathisia Rating Scale (BARS) | Baseline Day 1 to Week 52
  BARS is a 4-item rating scale used to assess drug-induced akathisia. The scale comprises items for rating the observable restless movements that characterize the condition, the subjective awareness of restlessness, and any distress associated with the akathisia (each on a 4-point scale from normal [0] to severe [3]). In addition, there is a global severity for akathisia rated on a 6-point scale (absent [0] to severe akathisia [5]).
Change From Baseline in Simpson-Angus Scale (SAS) | Baseline Day 1 to Week 52
  SAS is a 10-item rating scale for assessment of antipsychotic-induced parkinsonism in both clinical practice and research settings. Each item ranges from 0 (normal) to 4 (extreme symptoms). The scale consists of 1 item measuring gait (hypokinesia), 6 items measuring rigidity, and 3 items measuring glabella tap, tremor, and salivation, respectively.
Number of Participants With Clinically Significant Changes From Baseline in Opthalmologic Parameters | Baseline Day 1 to Week 52
  Ocular examination parameters included Intraocular pressure (IOP) measurement, Best-corrected visual acuity (BCVA), color fundus photography, color vision testing using Hardy Rand and Rittler (HRR) plates, and assessment of Optical coherence tomography (OCT) and cataracts. The investigator assessed the results for clinical significance.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (42):
- United States (40):
  - Harmonex Neuroscience Research /ID# 234938, Dothan, Alabama
  - Pillar Clinical Research /ID# 236434, Bentonville, Arkansas
  - Advanced Research Center /ID# 241903, Anaheim, California
  - Duplicate_Alliance for Research - Long Beach /ID# 236261, Long Beach, California
  - CHOC Children's Hospital /ID# 251019, Orange, California
  - ATP Clinical Research- Orange /ID# 257095, Orange, California
  - Prospective Research Innovations Inc /ID# 236098, Rancho Cucamonga, California
  - University of California, San Diego Department of Psychiatry /ID# 236466, San Diego, California
  - Pacific Clinical Research Management Group /ID# 234377, Upland, California
  - D&H Doral Research Center-Doral /ID# 255459, Doral, Florida
  - Sarkis Clinical Trials /ID# 236893, Gainesville, Florida
  - Galiz Research- Palmetto Medical Plaza /ID# 236277, Hialeah, Florida
  - Advanced Research Institute of Miami /ID# 242505, Homestead, Florida
  - Duplicate_Sandhill Research LLC /ID# 251239, Lake Mary, Florida
  - Columbus Clinical Services, Llc /Id# 234281, Miami, Florida
  - G+C Research Group, LLC /ID# 261398, Miami, Florida
  - Florida Research Center, Inc. /ID# 236515, Miami, Florida
  - Links Clinical Trials /ID# 240975, Miami, Florida
  - South Florida Research Ph I-IV /ID# 237453, Miami Springs, Florida
  - K2 Medical Research - Orlando - South Orlando Avenue /ID# 257528, Orlando, Florida
  - APG Research, LLC /ID# 251153, Orlando, Florida
  - D&H Tamarac Research Center /ID# 250435, Tamarac, Florida
  - Atlanta Center for Medical Research /ID# 234698, Atlanta, Georgia
  - CenExcel iResearch LLC /ID# 237391, Decatur, Georgia
  - Atlanta Behavioral Research, LLC /ID# 236374, Dunwoody, Georgia
  - Ascension Illinois /ID# 235857, Hoffman Estates, Illinois
  - Med Clinical Research Partners LLC /ID# 236071, Irvington, New Jersey
  - Erie County Medical Center /ID# 237204, Buffalo, New York
  - New Dawn Psychiatric Services PLLC /ID# 236597, Kinston, North Carolina
  - Quest Therapeutics of Avon Lake /ID# 235956, Avon Lake, Ohio
  - University of Cincinnati /ID# 236913, Cincinnati, Ohio
  - Cincinnati Children's Hospital /ID# 251020, Cincinnati, Ohio
  - CincyScience /ID# 236390, West Chester, Ohio
  - Cutting Edge Research Group /ID# 236664, Oklahoma City, Oklahoma
  - BioBehavioral Research of Austin /ID# 236479, Austin, Texas
  - Cedar Health Research /ID# 259364, Dallas, Texas
  - Red Oak Psychiatry Associates /ID# 236602, Houston, Texas
  - AIM Trials /ID# 236368, Plano, Texas
  - Family Psychiatry of The Woodlands /ID# 236426, The Woodlands, Texas
  - Core Clinical Research /ID# 236409, Everett, Washington
- Puerto Rico (2):
  - Dr. Samuel Sanchez PSC /ID# 246047, Caguas
  - GCM Medical Group PSC /ID# 246048, San Juan

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — http://www.abbvieclinicaltrials.com/study/?id=3070-301-001